CLINICAL TRIAL: NCT01197079
Title: Perception, Awareness, and Acceptance of Human Papillomavirus Disease and Vaccine Among Parents of Boys Aged 9 to 18 Years
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Tina Q. Tan, Professor of Pediatrics, Attending Physician - Infectious Diseases, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: Merck IISP 37875
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Human Papillomavirus (HPV)
Keywords: HPV; Vaccine; Vaccine utilization; Disease awareness
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents - Private Pediatric Offices: Parents of Boys aged 9 to 18 years from Private Pediatric Offices
  Interventions: Other: Survey
- Parents - Public Health Clinics: Parents of Boys aged 9 to 18 years from Public Health Clinics

INTERVENTIONS:
Other: Survey — Self administered anonymous survey
  Groups: Parents - Private Pediatric Offices

SUMMARY:
The objectives of this study are:

1. to determine the degree of understanding and perceived risks for human papillomavirus (HPV) disease, to examine and assess attitudes for personal use of HPV vaccine and identify potential barriers to HPV vaccine access and utilization in a population of young men who have sex with men (MSM) (under 26 years of age)and in parents of boys aged 9 to 18 years
2. to determine HPV vaccine acceptance and predictors of acceptance in a population of young MSM and in patients of boys ages 9 to 18 years
3. to develop strategies to overcome potential barriers to vaccination and improve vaccine access and utilization via development of targeted educational initiatives.

ELIGIBILITY:
Inclusion Criteria:

* MSM group - under age 26 years
* Parent group - parent of boy(s) ages 9 to 18 years

Exclusion Criteria:

* MSM group - previous receipt of HPV vaccine
* Parent group - previous receipt of HPV vaccine by male child

Ages: 9 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young men who have sex with men (MSM) that obtain medical care from a Gay/Lesbian/Bisexual/Transgender community health clinic
  Parents of boys aged 9 to 18 years who obtain their medical care from several public health clinics or who obtain their medical care from private pediatrician offices in Chicago
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pediatric Private practice, Chicago, Illinois
  - Children's Memorial Hospital Uptown Clinic, Chicago, Illinois
  - Pediatric Private Practice, Chicago, Illinois
  - Erie Family Health Clinic, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Private pediatric practice, Evanston, Illinois
  - Pediatric Private practice, Evanston, Illinois